CLINICAL TRIAL: NCT02800499
Title: Domestic COPD Patients Registry Business and COPD Phenotype Research Based by Registry Data - Multi-centered Trial
Brief Title: KOrea COpd Subgroup Registry and Subtype Research
Acronym: KOCOSS
Status: Enrolling by invitation | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Kwang-Ha Yoo, Professor, Konkuk University Medical Center
Other Study IDs: KUH1010338
Record Dates: First submitted 2016-06-04; First posted 2016-06-15 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- KOCOSS: The KOrea COpd Subgroup Study team (KOCOSS) cohort is an ongoing, longitudinal, prospective, non-interventional observational study within the Korean COPD patients

SUMMARY:
The KOrea COpd Subgroup Study team (KOCOSS) cohort is an ongoing, longitudinal, prospective, non-interventional and observational study within the Korean COPD patients. The prevalence of early COPD (mild to moderate COPD based by 2011 GOLD(the Global Initiative for Chronic Obstructive Lung Disease) guideline) is high in Korea. However, the patients with early COPD are not underdiagnosed due to mild symptom. The purpose of this study is to investigate early COPD characteristics and disease course and to form a guideline for early detection of COPD patients and prevention of progression to severe COPD.

DETAILED DESCRIPTION:
This study is a multicentered, observational study of the patients with COPD who were enrolled in 45 tertiary and university-affiliated hospitals from December 2012 to now.

The initial evaluation for all patients includes pulmonary function tests (PFT), 6-min walk distance (6MWD), COPD Assessment Test (CAT), modified Medical Research Council (mMRC) dyspnea scale, and the COPD-specific version of St. George's Respiratory Questionnaire (SGRQ-C), exacerbations in the previous 12 months, smoking status, patient-reported education level, medications and comorbidities.

Pulmonary function tests (PFTs) are performed every 6 months and CAT, mMRC and SGRQ-C are evaluated every 6 months and 6 min walt test is performed every years during the whole period of study.

All of the data were reported using case-report forms (CRFs) which are completed by physicians or trained nurses, and the patients are to be evaluated at regular 6-month intervals after the initial examination.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years old South Korean COPD patients(Bronchodilator test results FEV1/FVC <0.7)
* COPD patients who complain of cough, sputum, dyspnea
* Unrelated smoking history

Exclusion Criteria:

* other disease like asthma patients which is similar to COPD symptoms.
* patients who is not suitable for pulmonary function test and communication
* myocardial infarction or cerebrovascular event within the previous 3 months
* pregnants
* patients who disagree with registration
* rheumatoid patients
* cancer patients(including metastatic cancer, leukemia, lymphoma)
* irritable bowel syndrome
* patients who use systemic steroids over 8 weeks due to other diseases except COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Disease(COPD)
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2042-02 (Estimated); Study Completion 2042-02 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbation | 5 years
  Number of events

SECONDARY OUTCOMES:
Pulmonary function tests | 5 years
  COPD severity will be assessed based on post-bronchodilator Forced expiratory volume in one second(FEV) and FEV1/FVC(Forced vital capacity). FEV1 to forced vital capacity (FVC) :Mild - FEV1/FVC<0.7, FEV1 ≥80% normal Moderate - FEV1/FVC<0.7, FEV1 50-79% normal; Severe - FEV1/FVC<0.70, FEV1 30-49% normal; Very Severe - FEV1/FVC<0.70, FEV1 <30% predicted. We will measure spirometry at screening and every 6 months.
Modified Medical Research Council [mMRC] dyspnea scale | 5 years
  mMRC dyspnea scale is five-point scale with higher scores indicating more severe dyspnea. We will assess mMRC at screening and every 6 months.
COPD Assessment Test (CAT) | 5 years
  The CAT score was also used for evaluation of dyspnea. It consists of 8 items, each scored from 0 to 5, with higher scores indicating a more severe symptom.We will measure CAT at screening and every 6 months.
6-min walk distance (6MWD) | 5 years
  The 6MWD has been used as a simple tool to assess overall exercise tolerance in COPD patients. We will measure 6 min walk distance by ATS guideline at screening and every 6 months during the follow-up period
the COPD-specific version of St. George's Respiratory Questionnaire (SGRQ-C) | 5 years
  to assess the health status from the patient's perspective .The SGRQ-C is a 14-item questionnaire that can be summarized as a total score, as well as by three component scores for symptoms, activities, and impacts. We will assess SGRQ at screening and every 6 months.
Percentage of Participants with smoking history | 5 years
  we will assess smoking history at screening and every 6 months
Percentage of Participants with Other Relevant Diseases | 5 years
  We will examine the relevant disease which is defined as respiratory diseases, cardiovascular diseases (ischaemic heart disease, heart failure, hypertension), and other diseases (osteoporosis, GERD(gastroesophageal reflux disease), hyperlipidemia, bronchiectasis, emphysema).
COPD Treatment | Through study completion, average 5 years
  COPD treatments are defined as inhaled therapies, oral therapies and other therapies administered during the enrollment and influenza vaccination and smoking cessation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Seok NA Jung, Doctor, Principal Investigator — Hallym University Medical Center
Locations (1):
- Konkuk University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fromer L, Cooper CB. A review of the GOLD guidelines for the diagnosis and treatment of patients with COPD. Int J Clin Pract. 2008 Aug;62(8):1219-36. doi: 10.1111/j.1742-1241.2008.01807.x. Epub 2008 Jun 28. PMID 18547365
- [Background] Department of Health. Our health, our lives our say. London: Department of Health 2006.
- [Background] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Background] Yoo KH, Kim YS, Sheen SS, Park JH, Hwang YI, Kim SH, Yoon HI, Lim SC, Park JY, Park SJ, Seo KH, Kim KU, Oh YM, Lee NY, Kim JS, Oh KW, Kim YT, Park IW, Lee SD, Kim SK, Kim YK, Han SK. Prevalence of chronic obstructive pulmonary disease in Korea: the fourth Korean National Health and Nutrition Examination Survey, 2008. Respirology. 2011 May;16(4):659-65. doi: 10.1111/j.1440-1843.2011.01951.x. PMID 21342331
- [Background] Bednarek M, Maciejewski J, Wozniak M, Kuca P, Zielinski J. Prevalence, severity and underdiagnosis of COPD in the primary care setting. Thorax. 2008 May;63(5):402-7. doi: 10.1136/thx.2007.085456. Epub 2008 Jan 30. PMID 18234906
- [Background] Mannino DM, Sonia Buist A, Vollmer WM. Chronic obstructive pulmonary disease in the older adult: what defines abnormal lung function? Thorax. 2007 Mar;62(3):237-41. doi: 10.1136/thx.2006.068379. Epub 2006 Nov 7. PMID 17090573
- [Background] Mannino DM, Doherty DE, Sonia Buist A. Global Initiative on Obstructive Lung Disease (GOLD) classification of lung disease and mortality: findings from the Atherosclerosis Risk in Communities (ARIC) study. Respir Med. 2006 Jan;100(1):115-22. doi: 10.1016/j.rmed.2005.03.035. PMID 15893923